CLINICAL TRIAL: NCT01321645
Title: Efficacy of Lesser Known Homoeopathic Medicines in Acne Vulgaris - Azadirachta Indica
Brief Title: Efficacy of Azadirachta Indica (Homoeopathic Medicine) in Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Miglani, Anjali (Individual)
Collaborators: Department of Indian Systems of Medicine and Homeopathy (Other)
Responsible Party: Principal Investigator, Dr. Anjali Miglani, Senior Medical Officer, Miglani, Anjali
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Acne-003
Record Dates: First submitted 2011-03-20; First posted 2011-03-23 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-10

CONDITIONS: Acne Vulgaris
Keywords: Acne Vulgaris; Homoeopathy; Homeopathy; Azadirachta Indica
MeSH Terms: conditions — Acne Vulgaris | interventions — neem oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Azadirachta Indica — To start with subjects will be prescribed Azadirachta Indica in 6 potency to be taken in form of pills 4 times a day for seven days. Dosage and frequency will be changed, if required, based on the condition of subject and their response according to homoeopathic principles.

SUMMARY:
Acne is one of the most common skin problems in teenagers and adolescents. There are many lesser known homoeopathic medicines which have been mentioned in the literature for treatment of acne but their potential has not been properly assessed /documented and therefore these medicines don't form a part of many prescriptions. As a part of this study,efficacy of Azadirachta Indica will be studied in the treatment of Acne vulgaris

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 12 to 25 years of age
* Presence of inflammatory and non-inflammatory lesions
* Able to follow-up according to protocol
* Patients not taking any medication for treatment of Acne in preceding one month.

Exclusion Criteria:

* Acne Conglobata
* Pregnant or Breast feeding females or females having intention of becoming pregnant
* Significant systemic disease
* Any drug/ alcohol addiction
* History of chronic diseases treated with medications in the preceding month which might affect acne condition and treatment outcome

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2011-03; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
percent change in acne lesion counts from the Baseline | 6 months

SECONDARY OUTCOMES:
change in quality of life of subjects from baseline | 6 months
  Change in Quality of life will be assessed based on Quality of Life Questionnaire to be filled by subjects at the start of Treatment and at the end of time frame.

CONTACTS AND LOCATIONS:
Overall Officials: Anjali Miglani, BHMS, Principal Investigator — Department of Indian Systems of Medicine and Homeopathy
Locations (1):
- Delhi Government Health Centre - Homoeopathic Dispensary - Sector 12, Dwarka, New Delhi, National Capital Territory of Delhi, India